CLINICAL TRIAL: NCT06487338
Title: Effect of Low-level Laser Therapy Versus Shock Wave Therapy on Pain and Function in Patients With Chronic Non-specific Low Back Pain: a Randomized Controlled Clinical Trial
Brief Title: Effect of Low-level Laser Therapy Versus Shock Wave Therapy on Pain and Function in Patients With Chronic Non-specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Hosam Magdy Metwally, Lecturer of physical therapy for neurology, October 6 University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2024
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2024-07

CONDITIONS: Low Back Pain
Keywords: Low-level laser therapy; Shock wave therapy; Pain; Function; Chronic Non-Specific Low Back Pain
MeSH Terms: conditions — Low Back Pain; Pain | interventions — Low-Level Light Therapy; Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Twenty patients will receive low-level laser therapy 3 times per week for a month
  Interventions: Other: Low-level laser therapy
- Group B (Experimental): Twenty patients will receive shock wave therapy 3 times per week for a month
  Interventions: Other: Shock wave Therapy

INTERVENTIONS:
Other: Low-level laser therapy — Is a form of medicine that applies low-level (low-power) lasers that relieve pain.The effects appear to be limited to a specified set of wavelengths
  Arms: Group A
Other: Shock wave Therapy — is a non-invasive treatment that stimulates the body's natural healing process. It can relieve pain and promote healing of injured tendons, ligaments, and other soft tissues
  Arms: Group B

SUMMARY:
A significant global source of disability is low back pain. Maladaptive variations in the level of activity in the lumbar musculature are one thing that could possibly contribute to persistent pain.

ELIGIBILITY:
Inclusion Criteria:

1. All patients will suffer from mechanical low back pain
2. Age will range from 20 to 40 years
3. All patients will have BMI range from 20-24

Exclusion Criteria:

1. History of radicular pain
2. Lumbar disc prolapse.
3. Visual problems
4. History of previous lumbar surgery
5. BMI more than 24

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-08-25 (Actual); Primary Completion 2024-10-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Oswestry low back disability questionnaire | 30 minutes
  The Oswestry Disability Index (also known as the Oswestry Low Back Pain Disability Questionnaire) is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome toolsFor each section the total possible score is 5: if the first statement is marked the section score = 0; if the last statement is marked, it = 5. If all 10 sections are completed the score is calculated as follows: Example: 16 (total scored) 50 (total possible score) x 100 = 32%
  If one section is missed or not applicable the score is calculated:
  16 (total scored) 45 (total possible score) x 100 = 35.5% Minimum detectable change (90% confidence): 10% points (change of less than this may be attributable to error in the measurement)
Back pain functional scale | 20 minutes
  The Back Pain Functional Scale (BPFS) is a subjective scale used to measure the patient's physical function after low back painThis scale consists of a total score of 60. Moreover, the patient's score can be measured from the responses obtained on the Likert scale (0 to 5), and accordingly, a total score is summed up out of 60. Furthermore, the maximum score obtained indicates the maximum physical abilities of the patients. In addition, this scale also has an 'Adjusted score' ranging from 0 (0%)-unable to perform any activity to 60 (100%)-no difficulty in any activity
Visual analogue scale | 5 minutes
  Visual analogue scale (VAS) is a unidimensional measure of pain intensity, used to record patients' pain progression, or compare pain severity between patients with similar conditions.
  Visual analogue scale (VAS) is most commonly a straight 100-mm line, without demarcation, that has the words "no pain" at the left-most end and "worst pain imaginable" (or something similar) at the right-most end.48 Patients are instructed to place a mark on the line indicating the amount of pain that they feel at the time of the evaluation. The distance of this mark from the left end is then measured, and this number is used as a numeric representation of the severity of the patient's pain

CONTACTS AND LOCATIONS:
Locations (1):
- October 6 University, Giza, Egypt